CLINICAL TRIAL: NCT02958007
Title: Peer Support for Exercise in Older Veterans With Psychotic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2339-W; 1IK2RX002339-01A1 (NIH)
Record Dates: First submitted 2016-11-02; First posted 2016-11-08 (Estimated); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2022-11

CONDITIONS: Psychotic Disorder
MeSH Terms: conditions — Psychotic Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peer Education on Exercise for Recovery (Experimental): A 24-week group-based peer coaching intervention delivered by a VA Peer Specialist, to promote participation in a supervised fitness training program and general physical activity
  Interventions: Behavioral: Peer Education on Exercise for Recovery
- Enhanced supervised fitness training (Active Comparator): A 24-week intervention to promote participation in a supervised fitness training program and general physical activity, which includes individual support from non-peer staff
  Interventions: Behavioral: Enhanced supervised fitness training

INTERVENTIONS:
Behavioral: Peer Education on Exercise for Recovery — A 24-week group-based peer coaching intervention delivered by a VA Peer Specialist, to promote participation in a supervised fitness training program and general physical activity
  Arms: Peer Education on Exercise for Recovery
Behavioral: Enhanced supervised fitness training — A 24-week intervention to promote participation in a supervised fitness training program and general physical activity, which includes individual support from non-peer staff
  Arms: Enhanced supervised fitness training

SUMMARY:
Older adults with psychotic disorders experience a dual set of challenges: those related to serious mental illness, and those related to aging. They have medical, cognitive, psychological and social difficulties; as a result they have an almost four times greater likelihood of early institutionalization in nursing homes. These challenges make it difficult for this group to engage in health behaviors, such as exercise. This is unfortunate, since participation in health-promoting activities is essential for maintaining functional independence with age. This study aims to develop and pilot test a peer coaching intervention for older Veterans with psychotic disorders, in which VA Peer Specialists, who are Veterans in recovery from mental illness, will provide intensive coaching to older Veterans with psychotic disorders to promote their participation in exercise and physical activity. Results from this study will inform us as to whether this intervention is acceptable to Veterans, feasible to implement, and effective in increasing exercise, physical activity, and physical fitness/function.

DETAILED DESCRIPTION:
Project was modified to minimize risk of exposure to COVID-19. Sample size was reduced due to loss of time due to pandemic restrictions.

Anticipated Impacts on Veteran's Healthcare: Older Veterans with psychotic disorders face unique barriers to engagement in health-promoting activities, including prototypical features of psychosis (e.g., negative symptoms, medication side effects) and exacerbating features of the aging process (e.g., increased medical comorbidity, declines in musculoskeletal health). It is critical to develop strategies to empower this group to overcome these barriers and engage in health behaviors that can improve their functioning and quality of life. Peer interventions, or interventions delivered by individuals who are similar to a patient population on some characteristic such as age or diagnosis, effectively promote engagement in health behaviors in a range of populations. Despite the promise of peer support and urgent needs of older adults with psychosis, there are no well-specified peer support interventions that promote participation in health behaviors and are tailored to the needs of this group. The present study will yield a well-specified group-based peer coaching intervention, to be delivered by VA Peer Specialists (Veterans in recovery from mental illness), targeted to empower older Veterans with psychosis to overcome barriers, increase exercise/physical activity, and improve functioning.

Project Background: Over the next two decades, Veterans with psychotic disorders (i.e., schizophrenia spectrum disorders and affective psychoses) will age into older adulthood in unprecedented numbers. The challenges of treating this growing population and associated high costs will have profound implications for VHA. Older adults with psychotic disorders exhibit diminished physical and psychosocial functioning and are at increased risk for rapid functional decline and early institutionalization in nursing homes. Participation in structured exercise delays functional disability in older adults; however, older adults with psychosis exhibit low exercise participation. While peer-delivered exercise interventions for older adults promote initiation and maintenance of exercise and physical activity, there are no peer-delivered exercise interventions tailored to the unique needs of older adults with psychosis. The present study aims to fill this critical gap.

Project Objectives: This study will develop and pilot test a well-specified, group-based peer coaching intervention tailored to the unique needs of older Veterans with psychotic disorders: Peer Education on Exercise for Recovery (PEER). PEER will provide intensive coaching from a VA Peer Specialist to promote participation in a supervised fitness training program for older Veterans. To develop the intervention, materials from existing peer-delivered wellness interventions for Veterans with serious mental illness will be tailored for older Veterans with psychosis, through an iterative process synthesizing the extant literature and pilot data, developing draft materials, and obtaining feedback from a multidisciplinary panel of expert mentors/consultants and Peer Specialists/Veteran consumers. A small open trial of PEER will be conducted with 6 older Veterans with psychotic disorders (ages 50 and up); qualitative interviews will explore participants' perceptions of PEER. Finally, a pilot randomized controlled trial (RCT) of PEER will be conducted. Older Veterans with psychotic disorders (ages 50 and up, n=22) will be enrolled in supervised fitness training and randomized to receive group-based peer coaching (the PEER condition) or individual support from non-peer staff (the enhanced supervised fitness training (ESFT) condition). Feasibility of PEER (rates of recruitment, intervention engagement, and peer coach fidelity) will be measured. The impact of PEER versus ESFT on attendance of exercise sessions, levels of physical activity, and physical functioning will be examined. Additionally, the PI will engage in training activities to develop expertise in the functional rehabilitation of older adults with psychosis.

Project Methods: This project will include developing intervention materials for PEER, conducting an open trial of PEER in a small sample, and completing a small RCT. The investigators will monitor acceptability and feasibility; study Veterans' experiences; and measure exercise/physical activity behaviors and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of a psychotic disorder, meeting criteria established by the VA Serious Mental Illness Treatment Research and Evaluation Center (SMITREC): schizophrenic disorders (295.0-295.9), affective psychoses (296.0-296.1, 296.4-296.8), or major depression with psychotic features (296.24, 296.34)
* age 50 or older
* participation in mental health services at the VA Maryland Healthcare System
* sufficient clinical stability to participate as deemed by a mental health treatment provider and/or chart review
* sufficient medical stability as deemed by a medical provider

Exclusion Criteria:

* Current participation in a supervised exercise program
* medical conditions which would preclude exercise participation including:

  * unstable angina
  * proliferative diabetic retinopathy
  * oxygen dependence
  * frank incontinence
  * open wounds
  * poorly controlled Type 2 diabetes (HbA1c > 9%)
  * current treatment for active cancer
  * New York Heart Association Stage II-IV heart failure
  * dialysis for chronic kidney disease
  * myocardial infarction in the previous three months
* problematic substance abuse/dependence
* imminent risk of suicidal or homicidal behavior
* lack of capacity to consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjana Muralidharan, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer Education on Exercise for Recovery | Enhanced Supervised Fitness Training
Started | 11 | 11
Completed | 10 | 8
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Education on Exercise for Recovery | Enhanced Supervised Fitness Training | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (4.1) | 64.4 (8.4) | 62.8 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Intervention Engagement
Description: Percent of participants randomized to PEER who attend at least three group sessions
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Peer Education on Exercise for Recovery
Number analyzed (Participants) | 11
Participants | 8

2. Primary Outcome: Intervention Fidelity
Description: Percent of sampled PEER group sessions in which the peer coaches were adequately adherent, as per the PEER Fidelity Measure. This measure includes content items (e.g., "How well did facilitators review the educational topic of the day") and process items (e.g., "How well did facilitators provide positive feedback and reinforcement throughout the class?") Each item is rated as 0 (unacceptable), 1 (acceptable), or 2 (excellent), and then an average score is calculated. Adequate adherence was defined as an average score of 1 or greater and no items rated as unacceptable.
Time Frame: 12 weeks
Population: 25% of recorded group sessions randomly selected and reviewed by independent rater for fidelity
Measure: Count of Units; unit: Recorded group sessions
Units Other Than Participants: Recorded group sessions
Arm/Group | Peer Education on Exercise for Recovery
Number analyzed (Participants) | 11
Number analyzed (Recorded group sessions) | 13
Recorded group sessions | 11

3. Primary Outcome: Attendance
Description: Attendance- mean number of supervised fitness training sessions attended
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Peer Education on Exercise for Recovery | Enhanced Supervised Fitness Training
Number analyzed (Participants) | 11 | 11
sessions | 11.8 (10.6) | 9.5 (7.1)
Statistical Analysis 1: Comparison: Peer Education on Exercise for Recovery vs Enhanced Supervised Fitness Training; Test type: Superiority; p = 0.544, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 weeks following randomization
Arm/Group | Peer Education on Exercise for Recovery | Enhanced Supervised Fitness Training
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/11
Other Adverse Events (participants affected / at risk) | 4/11 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Education on Exercise for Recovery (N=11) | Enhanced Supervised Fitness Training (N=11)
Acute hypoxic respiratory failure- unrelated to study (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — After randomization and prior to beginning fitness training, Veteran was admitted to hospital for acute encephalopathy, acute hypoxic respiratory failure and respiratory acidosis secondary to inhalant abuse. Veteran medically withdrawn from study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Education on Exercise for Recovery (N=11) | Enhanced Supervised Fitness Training (N=11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4)
Lightheaded during exercise (Nervous system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Fell in his home (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leg wound- unrelated to exercise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hernia- unrelated to study (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anxious distress at gym (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to COVID, this trial was shut down partway through for one year. The second half of the trial was conducted in a hybrid model, with all aspects of the study being conducted virtually except gym attendance. Due to this loss of time, the sample size was smaller than originally intended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT02958007/Prot_SAP_000.pdf